CLINICAL TRIAL: NCT06397586
Title: Effectiveness of Plyometric Training Based on Two Different Motor Imagery and Action Observation Tecniques Applied to Female Volleyball Players
Brief Title: Plyometric Training Based on Motor Imagery and Action Observation in Female Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ugur Cavlak (Other)
Collaborators: Biruni University (Other)
Responsible Party: Sponsor-Investigator, Ugur Cavlak, CLINICAL PROFESSOR, Biruni University
Organization: Biruni University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BiruniUnivi
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Motor Imagery
Keywords: Motor imagery; Plyometric Training; Dynamic Motor; Imagery; Volleyball
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP I: STATICK (Experimental): static motor imagery and movement observation-based plyometric training
  Interventions: Other: Routine volleyball
- GROUP II: DYNAMIC (Experimental): dynamic motor imagery and movement observation-based plyometric training
  Interventions: Other: Routine volleyball
- GROUP III: ACTIVE CONTROL (Active Comparator): plyometric training
  Interventions: Other: Routine volleyball

INTERVENTIONS:
Other: Routine volleyball — MOtor imagery
  Other Names: plyometric training

SUMMARY:
Plyometric training (PT) is training consisting of exercises that enable the muscles to reach maximum strength in minimum time. PE improves lower extremity muscle strength, jumping performance, agility, reaction time. Although plyometric exercises contribute greatly to increasing athlete performance, athletes cannot apply PE due to loading procedures at all times of the season. PEs in the literature generally involve active application of exercises. The definition of exercise includes not only physical exercise but also mental exercise. Athletes can use mental exercises as complementary training methods that can complement or add to physical training to compensate for their deficiencies. When mental exercises are examined, we often encounter two concepts. These are action observation (AO) and motor imagery (MI). MI imagines a task without actually performing it. AO is when a person watches a certain action being performed by another third party or while the video is being played back. There are studies showing that training on MI and AO methods creates more activation in the brain when applied together. Although the definition of motor imagery has been broadly separated from action, more recent imagery theories have led to the concept of dynamic motor imagery (DMI), the practice of athletes adopting a harmonious body position and embodying the spatial and temporal properties of movement without performing the entire movement. To the best of our knowledge, no study has been found in which PT based on MI and AO was performed on female volleyball players. Additionally, to our knowledge, the effectiveness of DMI on female volleyball players has not been investigated. Therefore, the aim of our study is; PT based on MI and AO is applied to female volleyball players in two different ways; The aim is to investigate the effects of balance, jumping, agility and reaction time and to compare the effectiveness of these two methods.

DETAILED DESCRIPTION:
45 licensed female volleyball players between the ages of 18 and 25 will be included in the study. Volleyball players will be randomized into three groups: Group A, Group B, Group C. Group A- Routine training + MI and AO; He/she will be included in an MI and AO based PT exercise program with a physiotherapist 2 days a week for 8 weeks. Group B- Routine training + DMI and AO will perform the same exercise program as DMI. Group C- Control group will continue their routine training program for 8 weeks. Demographic information of all patients to be included in the study will be recorded with the "Case Evaluation Form". The patients' static balances were measured with the Performanz device, their dynamic balances with the Y balance test, their jumping performances with the My Jump 2 application and one-step jump test, their agility performances with the shuttle running test and agility T test, their reaction times with the Blazepod device, their movement imagination abilities with the Movement Imagination Questionnaire. It will be evaluated with -3. All data will be evaluated using statistical analysis methods.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman between the ages of 18-25
* Becoming a licensed volleyball player
* Playing volleyball actively
* Knowing how to read and write Turkish to understand, interpret and answer surveys
* Having signed the informed consent form

Exclusion Criteria:

Athletes with acute injury and/or early postoperative surgery

* Those who suffered injuries while working
* Those who did not follow the research protocol (did not complete the tests and/or did not complete the training program)
* Those who want to leave the research voluntarily

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females Voleyball Olayers
Enrollment: 45 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Movement Imagination Questionnaire-3 | baseline and immediately after the intervention
  It was developed by Williams et al. and Dilek et al. in order to determine the imagination ability of all individuals included in the training and control groups. "Movement Imagination Questionnaire-3", whose Turkish validity and reliability has been established by , will be used (internal consistency coefficient: 0.87). With 12 items in this survey, internal visual imagery, external visual imagery and kinesthetic imagery abilities will be evaluated through four actions each. Actions will initially be taken actively by individuals. They were then asked to perform these actions as mental tasks. These mental tasks were scored using a seven-point Likert scale (1: very difficult to see and feel; 7: very easy to see and feel). In the score calculation, the score average of the four relevant actions will be taken for each of the three sub-dimensions
Vertical jump test | baseline and immediately after the intervention
  Vertical jump test will be used to determine the vertical jump distances of the participants. The jump test will be video recorded and analyzed with the help of the smartphone application "My Jump 2" (© 2016-18 Carlos Balsalobre-Fernández). It has been emphasized that there is a near-perfect similarity between the My Jump 2 application and the reactive force index, time on the ground and jump height measurements of the force platform, and therefore the application is a valid and reliable measurement method
Agility Performance Evaluation | baseline and immediately after the intervention
  Shuttle running test (MKT) is a test frequently used to evaluate agility in athletes. MKT test will be applied according to the recommendation of Leger and Lambert (1982). Running speed signals will be controlled with the Sportexpert Test Timer (Italy) pace generator device. The test will start at 8.5 km/h and increase by 0.5 km/h every minute. Participants were asked to travel 20m at each signal. The test will be terminated when the participants cannot complete the 20m distance three times in a row even though the signal sounds. The estimated VO2max values of the participants will be calculated with the formula suggested by Leger et al.
Agility T test | baseline and immediately after the intervention
  Agility T test consists of 4 contact points formed in a T shape in an area of 10m length and 10m width. The aim is to complete a series that requires the subject to move in different directions and in different ways between these contact points in the shortest time possible. The difference between this test and other agility tests is that the subject always looks in the same direction. It changes direction by sliding steps to the right and left or by running backwards. This test requires two 900° and 1800° turns, as well as 10m forward, 10m right, 10m left and 10m back, for a total distance of 40m
single-step hop test | baseline and immediately after the intervention
  The single-step hop test will be used, which has been found to have excellent test-retest reliability as an intraclass correlation coefficient of 0.94 for the dominant side and 0.96 for the non-dominant side

SECONDARY OUTCOMES:
Y balance test | baseline and immediately after the intervention
  Y balance test (YDT) will be used to evaluate dynamic balance. Measurement will be made with the "Y Balance Test" platform. YDT allows the participant to balance on one foot while simultaneously extending the other foot in three different directions as possible: anterior, posterolateral and posteromedial. The YDT composite score is calculated by summing the 3 reaching directions and dividing the results by the lower extremity length. YDT is one of the valid and reliable measurement methods used to evaluate balance in athletes
Static Balance test | baseline and immediately after the intervention
  Performance Balance system is an electronic monitoring device designed to analyze lower extremity muscle groups that affect human balance. The basic method used is to reveal the contraction behavior of the muscles by following the balance focus. The device will measure the differences between individuals' dynamic and static balance, eyes open and eyes closed balance, two-foot and single-foot (right/left) balance, and right/left foot balance, and first-test-last-test balance developments will be measured. During the test, the participant will be asked to stand on the balance system and maintain his balance by following the commands given. The platform is linked to computer software that allows the balance to be evaluated objectively. Thanks to this software, the researcher will be able to monitor the measurements from his tablet or laptop. Muscle structure and balance measurements of individuals will be evaluated according to the results of the balance tests
Evaluation of reaction time | baseline and immediately after the intervention
  Reaction times of the participants will be measured with the Blazepod (Israel) system, which consists of wireless light discs that can be controlled via an application compatible with smart devices. A validity and reliability study was conducted to evaluate the reaction time of the device (

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Scott M, Taylor S, Chesterton P, Vogt S, Eaves DL. Motor imagery during action observation increases eccentric hamstring force: an acute non-physical intervention. Disabil Rehabil. 2018 Jun;40(12):1443-1451. doi: 10.1080/09638288.2017.1300333. Epub 2017 Mar 21. PMID 28322596